CLINICAL TRIAL: NCT05040243
Title: A Randomized Controlled Double-blind Study of Acupuncture Combined With Yanqing Zhitong Ointment Acupoint Application in the Treatment of Chronic Non-specific Low Back Pain
Brief Title: Acupuncture Combined With Yanqing Zhitong Ointment Acupoint Application in Chronic Non-specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZYCCCX-1006
Record Dates: First submitted 2021-06-17; First posted 2021-09-10 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Non-specific Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): On the basis of conventional acupuncture treatment combined with acupoint application of Yanqing Zhitong Ointment.
  Acupuncture point:Weizhong,Shenshu,Dachangshu,Jaji,Ashi Acupoint application:Pain in the lumbar spine, Mingmen, Yaoyangguan, Shenshu (double), Ashi (6 points in total); Within 3 inches beside the spine on both sides of the waist, Shenshu (double), Dachangshu (double), Ashi (6 points in total); 3 inches away from the sides of the spine on both sides of the waist, Shenshu (double), Zhishi (double), Ashi (6 points in total).
  Stick to each point for about 4 hours. If there is a burning sensation or obvious itching or other discomfort on the part after application, it can be removed in advance.
  Three times a week( Monday, Wednesday, and Friday). Course of treatment: each course lasts for 2 weeks, a total of 2 courses of continuous treatment.
  Interventions: Other: Yanqing Zhitong Ointment Acupoint application
- Control Group (Sham Comparator): The control group was combined with placebo acupoint application on the basis of conventional acupuncture treatment.
  Placebo patch: colored and drug-free patch (composition: petrolatum, food coloring) Acupuncture, application of acupuncture points and treatment course were the same as those in the treatment group.
  Interventions: Other: placebo acupoint application

INTERVENTIONS:
Other: Yanqing Zhitong Ointment Acupoint application — Yanqing Zhitong Ointment is a traditional external preparation of experiential prescription, which is an extract made by water extraction and concentration of Qingfengteng, Corydalis yanhusuo, Interleukin, Kansui, Asarum, etc. Clinical studies in the past ten years have preliminarily shown that it has the effects of warming meridians, promoting blood circulation, dredging collaterals and relieving pain, and has a definite effect.
  Arms: Treatment Group
Other: placebo acupoint application — The control group was combined with placebo acupoint application on the basis of conventional acupuncture treatment.
  Placebo patch: colored and drug-free patch (composition: petrolatum, food coloring) Acupuncture, application of acupuncture points and treatment course were the same as those in the treatment group.
  Arms: Control Group

SUMMARY:
Carry out a randomized controlled double-blind study, the acupuncture combined with placebo application group was compared with the acupuncture combined with Yanqing Zhitong ointment acupoint application group, 86 patients with chronic non-specific low back pain were included.

DETAILED DESCRIPTION:
Treatment group(acupuncture combined with Yanqing Zhitong ointment acupoint sticking) Acupoints for manual acupuncture:Weizhong(BL40), Shenshu(BL23) ,Dachangshu(BL25) ,Geshu(BL17) ,Kunlun(BL60) ,Ashi point Acupoints for sticking:According to the location of pain, we select acupuncture points along the meridian

Controal group(acupuncture combined with placebo application) Interventions are same as Treatment Group.

Both groups were treated 3 times a week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic of non-specific low back pain
2. Aage from 18 to 65
3. Last for at least 12 weeks
4. VAS between 4 and 7
5. No other treatment in the past 3 months
6. Patients with no partial skin damage
7. No other relevant treatment methods
8. Sign informed consent and informed consent

Exclusion Criteria:

1. Pregnant women
2. Suffer from diabetes
3. With skin ulcers or contusion wounds
4. Past history of severe allergy to transdermal preparations
5. Complicated with serious diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Lumbar JOA Scale | Change from baseline JOA at 4weeks
  The JOA scale for low back pain consists of the patient's subjective symptoms (0-9 points), clinical signs (0-6 points), daily activity limitation (0-24 points) and bladder function (normal 0 points, slight loss of control-3 points, severe loss of control) -6 points) Four parts, a total score of 29 points. The total score reflects the symptoms and dysfunction of low back pain, and the score indicates the severity of the dysfunction.

SECONDARY OUTCOMES:
Lumbar JOA Scale | Change from baseline JOA at 2weeks and follow up 2weeks
  The JOA scale for low back pain consists of the patient's subjective symptoms (0-9 points), clinical signs (0-6 points), daily activity limitation (0-24 points) and bladder function (normal 0 points, slight loss of control-3 points, severe loss of control) -6 points) Four parts, a total score of 29 points. The total score reflects the symptoms and dysfunction of low back pain, and the score indicates the severity of the dysfunction.
Visual Analog Scoring (VAS) | Change from baseline VAS at 2weeks ,4 weeks and follow up 2weeks
  VAS is a pain scoring scale that is currently widely used in clinical practice. The scale uses a line segment or ruler with a length of 10 cm, and the subject makes corresponding marks on the line segment according to the subjective pain intensity.
Oswestry Dysfunction Index (ODI) | Change from baseline ODI at 2weeks ,4 weeks and follow up 2weeks
  ODI is a self-evaluation scale for dysfunction of patients with low back pain. It consists of 10 aspects including pain degree, personal living ability (washing, dressing), lifting, walking, sitting, standing, sleep influence, sex life, social activities and travel. Each aspect covers 6 options, with points ranging from 0 to 5 points. The lowest score indicates no abnormal dysfunction, and the highest score indicates severe dysfunction. The corresponding candidate content scores are added up in turn according to the scores, and the percentage of the total score in the highest score (50 points) of all content is obtained, which is called the Oswe-stry dysfunction index.
McGill Pain Questionnaire (MPQ) | Change from baseline MPQ at 2weeks ,4 weeks and follow up 2weeks
  MPQ is a multi-factor pain score scale, which establishes a three-dimensional structure of the nature of pain. MPQ has a higher evaluation dimension and can evaluate the multi-dimensional factors of pain. The higher the score, the more severe the pain.
Concise health scale SF-36 | Change from baseline SF-36 at 2weeks ,4 weeks and follow up 2weeks
  SF-36 is currently one of the most widely used universal health-related quality of life measurement tools in the world. SF-36 covers 8 dimensions for assessing health-related quality of life and a total of 36 content items. Each dimension includes: physical function (PF), role physical (RP), bodily pain (BP), General health (GH), vitality (VT), social function (SF), role-emotional (RE) and mental health (MH). SF-36 first calculates the original scores of the eight dimensions, and then obtains the final score after corresponding conversion. The final score is 0-100 points. The higher the final score, the better the health of the testee.
Tenderness threshold | Change from baseline tenderness threshold at 2weeks ,4 weeks and follow up 2weeks
  Use the digital pressure pain meter to measure the pressure pain threshold of soft tissues and muscles, and conduct an objective and quantitative assessment of pain. It is used for auxiliary diagnosis and scientific research of pain in muscles and tendons.
Averaged electromyography, AEMG | Change from baseline AEMG at 2weeks ,4 weeks and follow up 2weeks
  Surface electromyography (sEMG) is the bioelectric change of neuromuscular activity recorded from the surface of the muscle through electrodes, which can objectively reflect the activity level and functional state of the muscle. The electromyographic biofeedback meter was used to measure the surface electromyographic signals of the paraspinal muscles on both sides during the lumbar flexion and extension exercise in the standing position, and calculate the average electromyographic value (AEMG).

CONTACTS AND LOCATIONS:
Overall Officials: JIAN PEI, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital, Shanghai, China

REFERENCES:
- [Background] Maatta JH, Wadge S, MacGregor A, Karppinen J, Williams FM. ISSLS Prize Winner: Vertebral Endplate (Modic) Change is an Independent Risk Factor for Episodes of Severe and Disabling Low Back Pain. Spine (Phila Pa 1976). 2015 Aug 1;40(15):1187-93. doi: 10.1097/BRS.0000000000000937. PMID 25893353
- [Background] Garcia JB, Hernandez-Castro JJ, Nunez RG, Pazos MA, Aguirre JO, Jreige A, Delgado W, Serpentegui M, Berenguel M, Cantemir C. Prevalence of low back pain in Latin America: a systematic literature review. Pain Physician. 2014 Sep-Oct;17(5):379-91. PMID 25247896
- [Background] NIH Consensus Conference. Acupuncture. JAMA. 1998 Nov 4;280(17):1518-24. PMID 9809733
- [Background] Wen BL, Liu BY, Jin P, Wang XF, Xiang XX, Liu XF, Hu JQ, Lu F, He LY, Zhu WZ, Fang YG, Wang Y. Clinical research of acupoint application for "treatment of winter disease in summer" used to prevent and treat bronchial asthma in children. J Tradit Chin Med. 2012 Mar;32(1):31-9. PMID 22594099
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789